CLINICAL TRIAL: NCT03543592
Title: The Accuracy of Three-dimensional Power Doppler Ultrasound in the Diagnosis of Endometrial Lesions in Patients With Postmenopausal Bleeding Compared With the Endometrial Histopathology.
Brief Title: Three-dimensional Power Doppler in the Diagnosis of Endometrial Lesions in Patients With Postmenopausal Bleeding
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Cairo University (Other)
Responsible Party: Principal Investigator, Moutaz Sherbini, assistant professor, Cairo University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: 3081987
Record Dates: First submitted 2018-05-08; First posted 2018-06-01 (Actual); Last update posted 2020-05-19 (Actual); Status verified 2020-01

CONDITIONS: Postmenopausal Bleeding
Keywords: postmenopausal bleeding; ultrasound; power doppler; endometrium
MeSH Terms: interventions — Echocardiography, Doppler

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- 3 dimensional power Doppler (Other): 100 women suffering post-menopausal bleeding (occurred after at least 12 months of amenorrhea) will be included in the study and 3 dimensional ultrasonography and Doppler will be done for them
  Interventions: Diagnostic Test: 3 dimensional ultrasonography and Doppler

INTERVENTIONS:
Diagnostic Test: 3 dimensional ultrasonography and Doppler — Three-Dimensional images will be recorded. The volumes will be generated by the automatic rotation of the mechanical transducer 360 degrees. Visualization of the endometrium and myometrium in the three planes will be done to detect endometrial cavity and any lesions. The power Doppler gate will be activated for blood flow mapping of the endometrium and endometrial-myometrial interface (sub-endometrial area). The pulsed Doppler sample volume will be activated to obtain a flow velocity waveform (FVW). Vascularization index (VI), flow index (FI) and vascularization-flow index (VFI) will be automatically calculated from three consecutive FVWs.

SUMMARY:
100 women suffering post-menopausal bleeding will be included in the study. All the participants will undergo 3D Transvaginal Ultrasound to assess the endometrium and myometrium (for the presence of any focal lesions e.g. polypi) followed by 3D Power Doppler ultrasound assessment of the vascular indices: vascularization index (VI), flow index (FI) and vascularization-flow index (VFI) and endometrial volumes.

The results of the ultrasound and Doppler indices will be correlated to the histopathological examination of specimens collected following fractional curettage or hysterectomy.

DETAILED DESCRIPTION:
100 women suffering post-menopausal bleeding (occurred after at least 12 months of amenorrhea) will be included in the study.

After obtaining an informed consent entailing the explanation of the study and its aim, all participants will undergo the following; full history taking (including full menstrual history and the date of menopause), complete physical examination, laboratory investigations (complete blood count, liver function tests, kidney function tests and a coagulation profile). Baseline 2D transvaginal ultrasound will be done to measure endometrial thickness and to detect presence of any endometrial and myometrial focal lesions. 3D-transvaginal ultrasonography will be done to acquire multi-planner view of the uterine cavity and detect presence or absence of any cavitary or myometrial lesions and acquire endometrial volumes. This will be followed by 3D Power Doppler Ultrasound assessment of the vascular indices namely; vascularization index (VI), flow index (FI) and vascularization-flow index (VFI).

Transvaginal sonography will be performed for all patients using Voluson 730 PRO V transvaginal volumetric probe transducer with frequency range of 5-8 MHz equipped with color, power and pulsed Doppler capabilities. First, conventional gray-scale sonography will be performed to obtain longitudinal and transverse sections of the uterus. Maximum endometrial thickness (double-layer) will be measured in the longitudinal plane with the detection of any focal lesions.

For Three-Dimensional Ultrasound: Once the B - mode had been completed, three-dimensional images will be recorded. The volumes will be generated by the automatic rotation of the mechanical transducer 360 degrees. The probe will be kept steady, the patient will be asked to hold breath and volume mode will be switched on. With the use of the medium line density, the typical acquisition time will be between 4 and 10 seconds. Visualization of the endometrium in the three planes will be done to detect endometrial cavity. Endometrial margin, echogenicity and presence of intrauterine fluid will be examined to notice the presence of any heterogenic pattern, irregularity, asymmetry in the margin or local thickening denoting the presence of polyp, endometrial hyperplasia, or carcinoma. The myometrium will be also examined in the three planes to detect any other focal lesion e.g. Fibroid or Adenomyosis.

For Power Doppler Study, the power Doppler gate will be activated for blood flow mapping of the endometrium and endometrial-myometrial interface (sub-endometrial area). Power Doppler settings will be set to achieve maximum sensitivity for detecting low velocity flow without noise. Once the vessels have been identified, the pulsed Doppler sample volume will be activated to obtain a flow velocity waveform (FVW). Vascularization index (VI), flow index (FI) and vascularization-flow index (VFI) will be automatically calculated from three consecutive FVWs. Only endometrial and endometrial-myometrial interface vessels were included.

The patient will then be admitted for either a D and C operation (Endometrial curettage) or for Total Abdominal Hysterectomy. All removed tissues will be sent for histopathological examination of the endometrium or of any pathological uterine lesion. Pathological examination results will be correlated to ultrasound (2D and 3D) and Doppler findings,

ELIGIBILITY:
Inclusion Criteria:

• Post-menopausal bleeding (occurred after at least 12 months of amenorrhea)

Exclusion Criteria:

* History of hormone administration in the last 6 months.
* Systemic diseases causing abnormal uterine bleeding as hematologic diseases and chronic medical diseases.
* Women who experienced artificial or induced menopause because of the use of tamoxifen or any type of hormone replacement therapy.
* Patients who take any anticoagulant drugs.

Ages: 50 Years to 50 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 100 (Estimated)
Dates: Start 2018-06-01 (Actual); Primary Completion 2020-07-01 (Estimated); Study Completion 2020-08-15 (Estimated)

PRIMARY OUTCOMES:
the diagnostic performance of Vascularization index in detecting endometrial carcinoma | within 24 hours before the surgical procedure
  Vascularization index (VI) will be correlated to pathology report

SECONDARY OUTCOMES:
the diagnostic performance of the endometrial volumes acquired by Three-Dimensional Ultrasound | within 24 hours before the surgical procedure
  endometrial volumes will be correlated to pathology report
the diagnostic performance of flow index (FI) in detecting endometrial carcinoma. | within 24 hours before the surgical procedure
  flow index will be correlated to pathology report
the diagnostic performance of vascularization-flow index (VFI) in detecting endometrial carcinoma. | within 24 hours before the surgical procedure
  vascularization-flow index (VFI) will be correlated to pathology report

CONTACTS AND LOCATIONS:
Locations (1):
- kasr elaini hospital (Cairo university), Cairo, Egypt